CLINICAL TRIAL: NCT02375269
Title: A Randomized, Double- Blind Multicentric Study of the Effect of Remote Ischemic Preconditioning on Postoperative Complications in Patients Undergoing Major Minimal and Open Visceral Surgery
Brief Title: Effect of Remote Ischemic Preconditioning on Postoperative Complications in Visceral Surgery
Acronym: RIPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KEK-ZH-Nr. 2014-0458
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-01

CONDITIONS: Postoperative Complication
Keywords: Visceral Surgery; Comprehensive Complication Index; Patient undergoing abdominal surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIPC (Remote Ischemic Preconditioning) (Experimental): Preoperatively in the operation theater a tourniquet will be applied to the left arm and RIPC will performed. Therefore the tourniquet will be insufflated to suprasystolic pressure levels for 5 minutes, followed by 5 minutes reperfusion (deflated). Three cycles are planned. Duration of the procedure is 30 minutes.
  Interventions: Device: RIPC with a tourniquet
- Control (No Intervention): Preoperatively in the operation theater a tourniquet will be applied to the left arm. The tourniquet will not be insufflated. The tourniquet will be removed after 30 minutes.

INTERVENTIONS:
Device: RIPC with a tourniquet
  Arms: RIPC (Remote Ischemic Preconditioning)

SUMMARY:
Remote Ischemic Preconditioning (RIPC) is mediated by intermittent brief episodes (5-10 minutes) of short ischemia in a limb (i.e. arm), followed by reperfusion. For this purpose in 3-4 cycles, a tourniquet is insufflated to suprasystolic pressure levels for 5 minutes and deflated for 5 minutes afterwards. The ischemic episodes are known to stimulate platelets and factors platelet dependent factors such as Serotonin and VEGF. These humoral factors have a systemic effect and have the potential to protect target organs (i.e. heart, kidney, liver) remote to the ischemic limb.

The purpose of this randomized controlled study is to investigate the influence and impact of RIPC on postoperative complications in patients undergoing visceral surgery

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Undergoing major visceral surgery

Exclusion Criteria:

* < 18 years
* Pregnancy
* Signs of Infection/Inflammation on upper limb
* Shunt
* Medical history of axillary lymph node dissection
* Signs of malperfusion of upper limb (i.e. Allen Test)
* Missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications | 30 days
  Complications will be assessed by Comprehensive Complication Index and Dindo Clavien Score

SECONDARY OUTCOMES:
Hospital stay | 30 days
ICU stay | 30 days
Infection composite parameters | 30 days
  CRP, Procalcitonin, Leucocytes

CONTACTS AND LOCATIONS:
Overall Officials: Pierre- Alain Clavien, MD, Phd, Principal Investigator — Department of Surgery, Swiss HPB and Transplant Surgery, University Hospital Zurich, Switzerland
Locations (1):
- Department of Surgery, Swiss HPB and Transplant Surgery, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Oberkofler CE, Limani P, Jang JH, Rickenbacher A, Lehmann K, Raptis DA, Ungethuem U, Tian Y, Grabliauskaite K, Humar R, Graf R, Humar B, Clavien PA. Systemic protection through remote ischemic preconditioning is spread by platelet-dependent signaling in mice. Hepatology. 2014 Oct;60(4):1409-17. doi: 10.1002/hep.27089. Epub 2014 Aug 13. PMID 24700614
- [Background] Thielmann M, Kottenberg E, Kleinbongard P, Wendt D, Gedik N, Pasa S, Price V, Tsagakis K, Neuhauser M, Peters J, Jakob H, Heusch G. Cardioprotective and prognostic effects of remote ischaemic preconditioning in patients undergoing coronary artery bypass surgery: a single-centre randomised, double-blind, controlled trial. Lancet. 2013 Aug 17;382(9892):597-604. doi: 10.1016/S0140-6736(13)61450-6. PMID 23953384